CLINICAL TRIAL: NCT04615130
Title: Investigation of Outpatient PUlmonary REhabilitation in Patients Suffering From Post-PE Syndrome: a Randomized Waitlist-controlled Trial - the PURE-PE Study
Brief Title: PUlmonary REhabilitation in Patients Suffering From Post-PE Syndrome
Acronym: PURE-PE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stephan Nopp, Principal investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1335/2020
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Rehabilitation; Exercise Training; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: As the control group will undergo rehabilitation after the study period as well, it is possible to blind patients and outcome assessors to the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will undergo 6 weeks of outpatient rehabilitation.
  Interventions: Other: Rehabilitation
- Control (No Intervention): Patients will receive no intervention throughout the 6 weeks period.

INTERVENTIONS:
Other: Rehabilitation — Rehabilitation, exercise training
  Arms: Intervention

SUMMARY:
This study is a multicenter, parallel, randomized waitlist-controlled trial that primarily focuses on the short-term benefit of outpatient pulmonary rehabilitation (PR) on patients after acute pulmonary embolism.

Patients will be randomized into an intervention and a control group. The intervention group will receive 6 weeks of outpatient PR, while patients in the other treatment arm will serve as a control. After completion of the randomized study, the second arm will undergo PR as well.

ELIGIBILITY:
Inclusion Criteria:

* Post-PE syndrome (except patients previously diagnosed with CTEPH) diagnosed by any of the following:

  * Post-PE functional impairment criteria
  * Post-PE Cardiac Impairment criteria
  * Chronic Thromboembolic Disease criteria
* Possibility of starting rehabilitation between 12 and 36 weeks after the initial event of PE

Exclusion Criteria:

* CTEPH diagnosis
* Chronic pulmonary diseases: COPD, interstitial lung diseases, asthma (only patients with severe asthma defined as a FEV1 ≤ 80% will be excluded), a statement on COVID-19 was amended due to the pandemic #
* Active cancer
* Pregnancy
* Myocardial infarction or cardiac surgery one year prior to inclusion
* Congenital heart disease, congestive heart failure
* History of stroke
* Any previous inpatient or outpatient PR

Additional criteria that are absolute contraindications for pulmonary rehabilitation

* Acute and decompensated disease states with severe functional restrictions of various organ systems (e.g. heart, kidney and liver insufficiency, unstable angina pectoris, hemodynamically unstable arrhythmias, acute spinal cord injury, untreated hormonal disorders, acute psychological disorders)
* open tuberculosis
* active infectious diseases and acute inflammatory processes
* Stressful and time-consuming therapy that significantly impair the ability to rehabilitate (e.g. chemotherapy or radiation therapy after malignancy)
* Participants who are not sufficiently resilient due to physical or mental impairment and / or cannot be mobilized and therefore cannot actively use the rehabilitation facility
* lack of motivation for therapy
* massive incontinence
* drugs and alcohol addiction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walk Test | within the 6-week study period
  change of walking distance covered within 6 minutes before and after the intervention/control period, measured in meters

SECONDARY OUTCOMES:
peak oxygen consumption | within the 6-week study period
  change of peak oxygen uptake (VO2/kg/min) measured by lung spiroergometry
Maximal workload | within the 6-week study period
  change of maximal workload in cycle ergometer tests measured in Watt
One-repetition maximum for lower extremities | within the 6-week study period
  change of one-repetition maximum for lower extremities measured in kg
One-repetition maximum for upper extremities | within the 6-week study period
  change of one-repetition maximum for upper extremities measured in kg
Maximal inspiratory muscle pressure | within the 6-week study period
  change in maximum inspiratory muscle pressure measured in mbar
Inspiratory muscle endurance | within the 6-week study period
  change in inspiratory muscle endurance measured in seconds
Level of dyspnea | within the 6-week study period
  change in dyspea at rest and maximal exertion mesured with the medical research council scale and BORG scale
Health related quality of life | within the 6-week study period
  change of quality of life measured with the 5-level EQ-5D version (EQ-5D-5L)
Disease related quality of life | within the 6-week study period
  change of quality of life measured with the Pulmonary Embolism Quality of Life (PEmb-QoL)
Functional limitations | within the 6-week study period
  change of functional status measured with the patient reported outcomes measurement information system (PROMIS) physical function short form
Functional status | within the 6-week study period
  change of functional status measured with the post-VTE functional status scale (min: 0, max: 4, lower scores indicate better functional status)
Anxiety and depression | within the 6-week study period
  change in anxiety and depression measured with the hospital anxiety and depression scale (HADS)

CONTACTS AND LOCATIONS:
Locations (1):
- Therme Wien Med, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fabyan KD, Holley AB. Postpulmonary embolism syndrome. Curr Opin Pulm Med. 2021 Sep 1;27(5):335-341. doi: 10.1097/MCP.0000000000000789. PMID 34127618

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT04615130/Prot_SAP_002.pdf